CLINICAL TRIAL: NCT00102297
Title: A Phase 1 Study of the Safety, Pharmacokinetics, and Biologic Activity of Escalating Doses of FG-3019 in Subjects With Incipient Nephropathy Due to Type 1 or Type 2 Diabetes Mellitus
Brief Title: Study of the Safety of FG-3019 in Incipient Nephropathy Due to Type 1 or Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-MC3019-003
Record Dates: First submitted 2005-01-26; First posted 2005-01-27 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
Keywords: Incipient Nephropathy; Type 1 or Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — pamrevlumab

INTERVENTIONS:
Drug: FG-3019

SUMMARY:
The Phase 1b study is a multi-center trial designed to test the safety, tolerability, biologic activity of escalating doses of FG-3019 in up to 20 patients with type 1 or type 2 diabetes and microalbuminuria (early-stage kidney disease). Patients will receive either 3 or 10 mg/kg of FG-3019 administered every two weeks as an infusion for a total of four doses. The ability of FG-3019 to reduce the excretion of protein in the urine is being measured as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Body mass index not exceeding 32.0 kg/m2
* If female, subject must meet one of the following criteria: a) surgically sterile (hysterectomy or bilateral tubal ligation) OR b) at least two years postmenopausal OR c) using a dual method of contraception and have a negative serum pregnancy test if of childbearing potential
* Diagnosis of type 1 or type 2 diabetes according to the American Diabetes Association
* Fasting plasma glucose of ≥ 126 mg/dL or current treatment with oral hypoglycemic agents or insulin
* Microalbuminuria defined as albumin to creatinine ratio in a spot collection (first void) of 30 - 300 mg/gram confirmed by two samples two to three days apart
* Serum creatinine of no more than 1.5 mg/dL for men and no more than 1.1 mg/dL for women

Exclusion Criteria:

* Female subjects who are pregnant or lactating
* Non-diabetic renal disease
* History of allergic or anaphylactic reaction to human, humanized, chimeric, or murine monoclonal antibodies
* Coronary artery bypass graft surgery, myocardial infarction, cerebrovascular accident, percutaneous transluminal angioplasty, transient ischemic attack, history of unstable angina, known heart failure, uncontrolled cardiac arrhythmia, or uncontrolled hypertension within six months prior to Day 0
* Bilirubin, aspartate aminotransferase (AST), or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal
* History of cancer of any type in the past 5 years, except non- melanomatous skin cancer, localized bladder cancer, or in situ cervical cancer.
* Clinically significant and uncontrolled medical condition considered a high risk for participation in an investigational study
* Trauma or surgical procedures (including dental) within six months prior to Day 0
* Planned elective surgery during the study and for 3 months following the end of the study
* Participation in studies of investigational drugs within 6 weeks prior to first dose

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety
Tolerability
Pharmacokinetics

SECONDARY OUTCOMES:
Bioactivity on urinary and plasma markers

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA - LA BioMed, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Radiant Research, Dallas, Texas
  - Diabetes & Glandular Disease, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia